CLINICAL TRIAL: NCT06596928
Title: A Clinical Trial to Evaluate the Efficacy of a Men's Supplement in Supporting Testosterone, Improving Cognitive Function, Mood, and Sexual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scale Media Inc (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20430
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sexual Function; Cognitive Functions; Testosterone
Keywords: Mood

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Supplement Group (Experimental): Participants in this group will receive the test supplement (Essential Elements T-Hero Platinum). The supplement contains ingredients aimed at supporting testosterone levels, including Shoden® Ashwagandha Root and Leaf Extract.
  Interventions: Dietary Supplement: Essential Elements T-Hero Platinum
- Placebo Group (Placebo Comparator): Participants in this group will receive a placebo containing rice flour in a vegetable cellulose capsule.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Essential Elements T-Hero Platinum — Participants will take two capsules daily for 90 days
  Arms: Test Supplement Group
Dietary Supplement: Placebo — Participants in the placebo group will take two placebo capsules daily for 90 days.
  Arms: Placebo Group

SUMMARY:
This randomized, triple-blind, placebo-controlled, hybrid trial aims to evaluate the efficacy of a men's supplement designed to increase testosterone levels and improve energy, cognition, and sexual function. The study will involve 50 male participants, with assessments carried out at Baseline, Day 45, and Day 90 through questionnaires and blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Male (biological at birth).
* Aged between 30-65.
* Generally healthy - do not live with any uncontrolled chronic disease such as diabetes or hypertension.
* Willing to provide blood draws during the study duration.
* Fitness/wellness enthusiast who has the same weekly exercise routine i.e. HIIT, strength training, or running >3 times per week.
* Self-reported concerns with energy levels, mood, and libido and sexual performance/adequacy.
* Willing to avoid medications, supplements, or vitamins aimed at increasing testosterone levels for the duration of the study.

Exclusion Criteria:

* Any pre-existing chronic conditions that would prevent participants from adhering to the protocol, including oncological and psychiatric disorders.
* Anyone with known severe allergic reactions requiring the use of an Epi-Pen.
* Unwilling to follow the study protocol.
* Currently experiencing significant symptoms of a mental disorder that might interfere with study participation (e.g., eating disorder, obsessive-compulsive disorder, posttraumatic stress syndrome, bipolar disorder).
* Current substance abuse disorder.
* Any medical condition that is unstable or uncontrolled.
* Has introduced any new prescription medication or supplements within the past 12 weeks that influence testosterone production.
* History of testicular or prostate cancer.
* Previously has undergone a vasectomy.
* Currently undergoing hormone replacement therapy (HRT)
* Currently taking performance-enhancing drugs.
* Anyone taking prescription blood pressure, immunosuppressants, sleeping aids, anti-seizure, and/or thyroid medications.
* Living in New York, Rhode Island, Hawaii, or Alaska.

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Free and Total Testosterone Levels | Baseline, Day 45, Day 90
  This study will measure the changes in free and total testosterone levels in male participants. Blood samples will be collected at Baseline, Day 45, and Day 90. The primary goal is to assess the effectiveness of the test supplement in increasing testosterone levels compared to the placebo group.

SECONDARY OUTCOMES:
Change in Cognitive Function, Mood, Energy, and Sexual Function | Baseline, Day 45, Day 90
  This study will assess self-reported changes in cognitive function, mood, energy levels, and sexual function. Participants will complete validated questionnaires, including the Profile of Mood States (POMS) questionnaire, at Baseline, Day 45, and Day 90. The goal is to evaluate improvements in these parameters and their correlation with increased testosterone levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No